CLINICAL TRIAL: NCT07127198
Title: Tolerance and Appetite Reduction of a Nutritional Solution With Intragastric Gelation Properties
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2405NR
Record Dates: First submitted 2025-06-06; First posted 2025-08-17 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Weight Management
Keywords: weight; drink
MeSH Terms: conditions — Body Weight | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Interventional Product 1 (Active Comparator): Protein & Fiber - Variant 1
  Interventions: Dietary Supplement: Beverage Variant 1 (low gelation properties)
- Interventional Product 2 (Active Comparator): Protein & Fiber - Variant 2
  Interventions: Dietary Supplement: Beverage Variant 2 (medium gelation properties)
- Interventional Product 3 (Active Comparator): Protein & Fiber - Variant 3
  Interventions: Dietary Supplement: Beverage Variant 3 (high gelation properties)
- Comparator (Placebo Comparator): Protein & Fiber
  Interventions: Other: Control group (no gelation property)

INTERVENTIONS:
Dietary Supplement: Beverage Variant 1 (low gelation properties) — The first interventional product for this study is a drink containing protein and fiber at a concentration 1. It will come in a ready to drink format for the participants.
  Arms: Interventional Product 1
Dietary Supplement: Beverage Variant 2 (medium gelation properties) — The first interventional product for this study is a drink containing protein and fiber at a concentration 2. It will come in a ready to drink format for the participants.
  Arms: Interventional Product 2
Dietary Supplement: Beverage Variant 3 (high gelation properties) — The first interventional product for this study is a drink containing protein and fiber at a concentration 3. It will come in a ready to drink format for the participants.
  Arms: Interventional Product 3
Other: Control group (no gelation property) — The control product for this study is a drink containing protein and fiber. It will come in a ready to drink format for the participants.
  Arms: Comparator

SUMMARY:
The physical properties of a food product, such as its gelling properties in the stomach can influence how full a person may feel after its consumption. Decreasing appetite feeling through consumption of such a product with a low energy content may contribute to weight management.

The study will assess if a drink with gelation properties in the stomach can reduce appetite and therefore contribute to weight management.

This is a single-center, double-blinded, 4 arm cross-over randomized controlled study looking to enroll 24 adult participants. The study will be performed at the Clinical Innovation Lab (CIL), Nestlé Research, Lausanne. Enrolled participants will have 4 visit days after the screening visit. They will consume one of the test products, or control at each visit and complete the study assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female aged 18-65 years old (inclusive)
2. Body Mass Index (BMI) 27 - 32kg/m2 (inclusive), measured and defined by the site
3. Self-reported stable body weight for the past 6 months prior to screening (defined as not having gained or lost more than 5% of body weight)
4. Comfortable using technology, such as a smartphone or laptop
5. Willing and able to understand and sign a written informed consent prior to study entry
6. Deemed able to comply with the requirements of the study protocol and consume study products by study nurse

Exclusion Criteria:

1. Currently or in the last 3 months, use of medications affecting weight, study outcomes, including fat absorption such as, but not limited to: GLP-1 receptor analogues, SGLT-2 inhibitors, weight loss medications, medications that affect gastric pH, and any of the following drugs: cephaloridine, verapamil, valproic acid, and sulfonylureas, usually acting by competitive inhibition of L-carnitine transport by OCTN2, Orlistat, antacids, proton pump inhibitors, antibiotics, steroids or medications affecting thyroid hormones or gut hormones, antipsychotic medications, or antidepressants. As reported by participant.
2. Diagnosed with Eating behaviour disorders such as emotional or restrained eating determined or any ongoing psychiatric illness. As reported by participant.
3. Currently or within the last 3 months or planning to during the course of the study being on a weight loss regime (defined by actively following a diet such as Atkins, weight watchers, meal replacements, low or very low carbohydrate diet, ketogenic diet, intermediate fasting or enrolled into a governmental health program) or applying significant restrictions on food intake (i.e., regular breakfast skipping, regular cut on carbohydrates, regular intermittent fasting, diet reducing a specific macronutrient, diet significantly reducing calorie intake, excluding a group of food that was not excluded before). As reported by participant.
4. Any known/suspected food allergies. As reported by participant.
5. Currently pregnant, lactating, or breastfeeding. As reported by participant.
6. Unstable diagnosed chronic conditions (such as hypertension, cardiovascular diseases, liver diseases, renal diseases, metabolic diseases). Unstable is defined as a change in medications in the past 3 months, or a change in disease severity in the past 3 months. As reported by participant.
7. Acute GI upset (such as diarrhoea/constipation in the last 2 weeks, abdominal cramping etc.). As reported by participant.
8. Diagnosed with chronic GI disorder such as inflammatory bowel disease, Crohn's disease, ulcerative colitis, or irritable bowel syndrome. As reported by participant.
9. Ever underwent surgery for weight loss such as bariatric procedures or gastric bypass. As reported by participant.
10. Recent blood donation (<8 weeks). As reported by participant.
11. Current or past smokers (stopped less than 3 months ago). As reported by participant.
12. Any drug abuse within the past year. As reported by participant.
13. Alcohol consumption above levels recommended for healthy adults: Average alcohol intake > 2 standard drinks per day over a week for males or > 1 standard drink per day over a week for females as reported by the participant. One standard drink contains 10-12 g of ethanol, i.e., 0.3 dl of strong alcohols, 1dl of wine, 3 dl of beer. As reported by participant.
14. Currently participating in another interventional study. As reported by participant.
15. Family or hierarchical relationships with the research team members. As reported by participant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2025-05-22 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Incremental Area Under the Curve (iAUC) of the composite appetite score (CAS) | Time frame used to assess product difference are -5, +15, +30, +45, +60, +90, +120 minutes post product intake. Time frame collection is -120, -90, -60, -30, -5, +15, +30, +45, +60, +90, +120min post product intake.
  Incremental Area Under the Curve (iAUC) of the composite appetite score (CAS) derived from a 100 mm visual analogue scale (VAS) questionnaire on appetite.

SECONDARY OUTCOMES:
Gastrointestinal (GI) smart questionnaire score | Time frame used to assess product difference is -5, +30, +60, +90 and +120 minutes post product intake. However, time frame for collection is -120, -60, -5, +30, +60, +90 and +120 minutes post product intake.
GI hormones (ghrelin, GLP-1, PYY, GIP, CCK) levels postprandial and quantity of an ad libitum meal consumption 2hs after product intake and throughout the rest of the day | 5 minutes before IP intake and 15, 30, 45, 60, 90 and 120 minutes after IP intake
iAUC of the composite appetite score (CAS) | From -120, -90, -60, -30, -5 minutes before IP consumption to +15, 30, 60, 90 and 120 minutes after IP consumption, at V1, V2, V3 and V4

OTHER OUTCOMES:
Blood insulin and blood amino acid levels | 5 minutes before IP intake and 15, 30, 45, 60, 90 and 120 minutes after IP intake
iCmax and Tmax of the CAS. | From -120, -90, -60, -30, -5 minutes before IP consumption to +15, 30, 60, 90 and 120 minutes after IP consumption, at V1, V2, V3 and V4
  0-120 min ICmax and Tmax of the postprandial CAS
Individual components of the composite VAS scores in response the 4 products | From -120 minutes before IP intake to +120 minutes after IP intake atV1, V2, V3 and V4

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Innovation Lab - Nestlé Research, Lausanne, Switzerland